CLINICAL TRIAL: NCT06952257
Title: Pilot Study: Relationship Between Anesthetic Regimen and Bone Cement Implantation Syndrome
Brief Title: Relationship Between Anesthetic Regimen and Bone Cement Implantation Syndrome (BCIS)
Acronym: BCIS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00462108
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Bone Cement Implantation Syndrome
Keywords: Bone Cement Implantation Syndrome; Hip fracture; Anesthesia
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Active Comparator): Patients undergoing cemented hemiarthroplasty under general anesthesia
  Interventions: Procedure: Administration of general anaesthesia
- Neuraxial Anesthesia (Active Comparator): Patients undergoing cemented hemiarthroplasty under neuraxial anesthesia
  Interventions: Procedure: Neuraxial Analgesia

INTERVENTIONS:
Procedure: Administration of general anaesthesia — The anaesthesia will be administered intravenously
  Arms: General Anesthesia
Procedure: Neuraxial Analgesia — Will be administered as an epidural
  Arms: Neuraxial Anesthesia

SUMMARY:
The annual incidence of geriatric hip fractures in the United States is 325,000 and is projected to rise given the aging population.1 The mainstay of treatment is cemented hip hemiarthroplasty. Bone cement implantation syndrome (BCIS) is a serious perioperative complication unique to cemented arthroplasty characterized by hypoxia, hypotension, cardiac arrhythmias, and in severe cases, cardiac arrest. BCIS is associated with significantly higher rates of unplanned intubation, vasopressor use, prolonged hospitalization, and 30-day mortality.

Given the rising incidence of hip fractures, the identification of readily modifiable risk factors for BCIS such as anesthetic regimen is crucial to reduce morbidity and mortality. However, a prospective study comparing the rate of BCIS development between general and neuraxial anesthesia is currently lacking. Additionally, no studies have examined how the anesthetic regimen affects histamine and complement levels. Therefore, this pilot study aims to investigate the effect of anesthetic regimen on BCIS development as well as on histamine and complement levels in patients undergoing cemented hemiarthroplasty for hip fracture. The investigators hypothesize that neuraxial anesthesia will be associated with lower rates of BCIS as well as lower histamine and complement levels compared to general anesthesia.

The primary objective of this pilot study is to compare the effect of general and neuraxial anesthesia on the incidence and severity of BCIS in patients undergoing cemented hemiarthroplasty for hip fracture.

Secondary objectives include examining postoperative outcomes associated with BCIS, such as cardiac arrhythmias, unplanned intubation, hypoxia necessitating supplemental oxygen, altered mental status, and in-hospital mortality.

Additional objectives include comparing histamine and complement levels between anesthetic regimens as well as between patients with and without BCIS

DETAILED DESCRIPTION:
This study will be a prospective, randomized pilot study involving adult patients undergoing cemented hemiarthroplasty for hip fracture within the Johns Hopkins healthcare system. In total, 20-24 participants will be randomly assigned to receive either general anesthesia or neuraxial anesthesia with sedation. The use of general or neuraxial anesthesia in this study is consistent with the current standard of care for hip hemiarthroplasty. Randomization will be performed via computer-generated sequences and allocation concealment will be maintained. Blinding patients, anesthesiologists, and orthopedic surgeons to the anesthetic regimen is not possible, but the investigator(s) conducting the statistical analyses will be blinded to the anesthesic regimen.

Patients presenting to the Johns Hopkins system with a hip fracture will be screened for possible participation. If eligible for inclusion, informed consent will be obtained from the patient preoperatively. Patients will subsequently undergo a cemented hip hemiarthroplasty with an orthopedic surgeon under either general or neuraxial anesthesia. Intraoperative vital signs will be monitored in standard fashion and used to detect development of BCIS based upon previously established criteria.

Histamine and complement levels will be measured via blood samples collected at three timepoints: pre-operation, post-induction of anesthesia, and post-cementation. The collection of these labs is for research purposes only and is not part of routine care. Postoperative complications within 30-days of the index surgery will be identified via chart review. Thus, the study duration is 30 days for each patient and requires one visit (hospitalization with index surgery).

Patients that are randomly assigned to neuraxial anesthesia but require conversion to general anesthesia due to unsuccessful spinal or epidural will be considered a treatment failure. These patients will be analyzed per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old that are indicated for cemented hemiarthroplasty for hip fracture.

Exclusion Criteria:

* Patients with medical comorbidities that preclude randomization to an anesthetic regimen (e.g., severe aortic stenosis contraindicating general anesthesia or therapeutic anticoagulation contraindicating neuraxial anesthesia) or
* a severe cognitive impairment that precludes the ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-04-16 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Hypoxia | Intra-operatively, approximately 10 minutes
  Grade 1 BCIS, defined as moderate intraoperative hypoxia (<94%) or drop in systolic blood pressure of >20%) intraoperatively.
  Grade 2 BCIS, defined as severe hypoxia (<88%) or drop in systolic hypotension >40%.
  Grade 3 BCIS, defined as cardiovascular collapse requiring cardiopulmonary resuscitation.

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure (mmHg) | Immediately before injection, int-operative up to 10 minutes
  Blood pressure will be monitored at two independent time points: (1) immediately before cement injection and (2) Intraoperative nadir after cement injection.
Oxygen Saturation | Immediately before injection, intr-operative up to 10 minutes
  Oxygen saturation will be monitored at two independent time points: (1) immediately before cement injection and (2) Intraoperative nadir after cement injection.

CONTACTS AND LOCATIONS:
Overall Officials: Adam S. Levin, MD, Principal Investigator — Johns Hopkins Hospital, Dept Orthopedic Surgery, Baltimore, MD 21287
Locations (1):
- Dept of Orthopadic Surgery, Johns Hopkins Hospital, JHOC 5221, 601 N. Caroline St., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zastrow RK, Rao SS, Morris CD, Levin AS. The Effect of Anesthetic Regimen on Bone Cement Implantation Syndrome in Cemented Hemiarthroplasty for Hip Fracture. J Am Acad Orthop Surg. 2025 Jan 1;33(1):e46-e57. doi: 10.5435/JAAOS-D-24-00239. Epub 2024 Aug 30. PMID 39231275
- [Background] Rao SS, Suresh KV, Margalit A, Morris CD, Levin AS. Regional or Neuraxial Anesthesia May Help Mitigate the Effects of Bone Cement Implantation Syndrome in Patients Undergoing Cemented Hip and Knee Arthroplasty for Oncologic Indications. J Am Acad Orthop Surg. 2022 Feb 1;30(3):e375-e383. doi: 10.5435/JAAOS-D-21-00553. PMID 34844261